CLINICAL TRIAL: NCT03804463
Title: The Randomized Multicentic Prospective Controlled Trial in Fertility-sparing Treatment and Ovarian Preservation Management for Early Endometrial Cancer
Brief Title: The Multicentic Trial in Fertility-sparing Treatment and Ovarian Preservation Management for Early Endometrial Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Wang (Other)
Collaborators: First Hospital of China Medical University (Other)
Responsible Party: Sponsor-Investigator, Min Wang, Director, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017PS017K
Record Dates: First submitted 2018-06-04; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Endometrial Cancer
Keywords: Preservation of fertility surger; ovarian preservation; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- radical surgery group (Experimental): Endometrial cancer radical surgery to be administered in this arm.
  Interventions: Procedure: endometrial cancer radical surgery
- fertility preservation group (Experimental): Fertility-sparing surgery to be administered in this arm.
  Interventions: Procedure: fertility-sparing surgery
- ovarian preservation group (Experimental): Ovarian preservation surgery to be administered in this arm.
  Interventions: Procedure: ovarian preservation surgery

INTERVENTIONS:
Procedure: endometrial cancer radical surgery — Take hysterectomy and bilateral adnexectomy.
  Arms: radical surgery group
Procedure: fertility-sparing surgery — Take endometrectomy , preserve uterus and bilateral ovaries.
  Arms: fertility preservation group
Procedure: ovarian preservation surgery — Take hysterectomy,preserve bilateral ovaries.
  Arms: ovarian preservation group

SUMMARY:
Through multicenter, prospective, randomized, controlled clinical studies comparing different treatment options (fertility-sparing surgery and ovarian preservation surgery and radical surgery)therapeutic efficacy, safety and quality of life of patients, exploration of the best strategies and risks for the treatment of early endometrial cancer, and promotion and application.

DETAILED DESCRIPTION:
Patients eligible for enrollment are selected and divided into three groups randomly, including fertility group,ovarian preservation group and endometrial cancer radical surgery group. Take interventions including fertility preservation surgery,ovarian preservation surgery and endometrial cancer radical surgery for patients in different groups respectively. Compare therapeutic efficacy, safety and quality of life of patients to evaluate three treatment and explore the best treatment for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women, age ≤ 50 years
2. Surgical curettage / hysteroscopic pathology confirmed, endometrioid adenocarcinoma G1/G2 (including well-differentiated, high-medium and middle-differentiation);
3. Clinical consideration of IA (<1/2 muscle infiltration);
4. First-time treatment
5. The subject (or his legal representative) must understand the nature of the study and sign an informed consent form.

Exclusion Criteria:

1. At the same time participate in other clinical trials;
2. Can not tolerate surgery;
3. Ovarian suspicious metastasis;
4. Have a family history of ovarian cancer;
5. Incorporate other malignant tumors;
6. Preoperative CA125 abnormal persons

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-01-10 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Total survival Time | 6 months
  calculate the time from patients enter the group to death

SECONDARY OUTCOMES:
the change of Ovarian volume | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  measure the ovarian volume dynamically by ultrasonography
the change of endocrine function evaluation | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  measure the endocrine function(hormone level) dynamically by blood detection
Progression Free Survival | 6 months
  calculate the time from patients enter the group to tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Min Wang, PHD., Study Director — Shengjing Hospital
Locations (1):
- Shengjing Hospitaol of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No